CLINICAL TRIAL: NCT05468762
Title: Ultrasound arteriaL Stiffness evaluatIon and vaScular Complications in Patients Undergoing Transfemoral tranScatheter Aortic valvE Implantation: ULISSE Study.
Acronym: ULISSE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Giuseppe Musumeci (Other)
Responsible Party: Sponsor-Investigator, Dr. Giuseppe Musumeci, Dr. Giuseppe Musumeci, Azienda Ospedaliera Ordine Mauriziano di Torino
Organization: Azienda Ospedaliera Ordine Mauriziano di Torino (Other)
Other Study IDs: ULISSE
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Transfemoral tranScatheter Aortic valvE Implantation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transfemoral tranScatheter aortic valvE implantation — Transcatheter aortic valve implantation (TAVI) is an established treatment modality in patients ≥ 75 years old with severe symptomatic aortic stenosis after Heart Team evaluation

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is an established treatment modality in patients ≥ 75 years old with severe symptomatic aortic stenosis after Heart Team evaluation (1). Patients with high/prohibitive surgical risk and life expectancy ≥ 1 years are candidates for TAVI according to the current guidelines (1). Nowadays is expected a progressive increase of TAVI procedures, in relationship to aging and increased life expectancy (2). Percutaneous, particularly trans-femoral, access represents the best choice in the vast majority of TAVI patients, because of its minimal invasiveness and reduced mortality, due to lower rates of periprocedural bleedings and strokes (3,4). Technical advancements, improving expertise and simplification of procedure, lead to reduction of vascular complications, still significant, and linked with worst patients' outcome (5). Some factors are considered to increase the risk of vascular complication: patient related and procedural related factors. Patient-related factors include female gender, severe vascular calcification and peripheral vascular disease. Procedural related risk factors consist of increased sheath to femoral artery ratio (SFAR) and TAVI centre experience/case load (5). Considering the last 10 years progress in techniques, devices technology and clinical outcome, a new Valve Academic Research Consortium (VARC) consensus manuscript was published to provide an update of these emerging clinical and research issues in aortic valve therapy (6).

Arterial stiffness is a physiologic phenomenon occurring with age and involving changes in extracellular matrix components of the arterial wall. Particularly, the elastin fibres undergo proteolytic degradation and chemical alteration, with consequent increased production of collagen, by vascular smooth muscle cells with progressive arterial wall stiffening (7). Arterial stiffness appears to be accelerated under pathological conditions, such as hypertension, smoking, diabetes mellitus (DM) and kidney disease (8), furthermore has been shown to have two-fold higher incidence in women compared to men (9).

TAVI patients have higher median age and comorbidities, directly correlated with arterial stiffness (7), and female gender is a considered high-risk feature for vascular complication independently from SFAR and atherosclerosis (5).

Arterial stiffness induces progressive reduction of tensile strength, elongation and burst pressure with consequent drop of vessels breakpoint (10), that could be associated with vascular complications. Particularly, femoral artery stiffness could predispose to microlesions formation at TAVI device access, inducing vascular closure devices failure and vascular complications. Furthermore, vessel rigidity can be associated with a higher resistance during TAVI device delivery and increased probability of vessels injury (especially in presence of tortuosity and small artery diameters). Nowadays, there are no studies evaluating the relationship between arterial stiffness and TAVI vascular complications.

The aim of this study is to evaluate the relationship between arterial stiffness and TAVI vascular complications, defining a new predictor of vascular complications in order to give more accurate information for procedures planning.

DETAILED DESCRIPTION:
Background Transcatheter aortic valve implantation (TAVI) is an established treatment modality in patients ≥ 75 years old with severe symptomatic aortic stenosis after Heart Team evaluation (1). Patients with high/prohibitive surgical risk and life expectancy ≥ 1 years are candidates for TAVI according to the current guidelines (1). Nowadays is expected a progressive increase of TAVI procedures, in relationship to aging and increased life expectancy (2). Percutaneous, particularly trans-femoral, access represents the best choice in the vast majority of TAVI patients, because of its minimal invasiveness and reduced mortality, due to lower rates of periprocedural bleedings and strokes (3,4). Technical advancements, improving expertise and simplification of procedure, lead to reduction of vascular complications, still significant, and linked with worst patients' outcome (5). Some factors are considered to increase the risk of vascular complication: patient related and procedural related factors. Patient-related factors include female gender, severe vascular calcification and peripheral vascular disease. Procedural related risk factors consist of increased sheath to femoral artery ratio (SFAR) and TAVI centre experience/case load (5). Considering the last 10 years progress in techniques, devices technology and clinical outcome, a new Valve Academic Research Consortium (VARC) consensus manuscript was published to provide an update of these emerging clinical and research issues in aortic valve therapy (6).

Arterial stiffness is a physiologic phenomenon occurring with age and involving changes in extracellular matrix components of the arterial wall. Particularly, the elastin fibres undergo proteolytic degradation and chemical alteration, with consequent increased production of collagen, by vascular smooth muscle cells with progressive arterial wall stiffening (7). Arterial stiffness appears to be accelerated under pathological conditions, such as hypertension, smoking, diabetes mellitus (DM) and kidney disease (8), furthermore has been shown to have two-fold higher incidence in women compared to men (9).

TAVI patients have higher median age and comorbidities, directly correlated with arterial stiffness (7), and female gender is a considered high-risk feature for vascular complication independently from SFAR and atherosclerosis (5).

Arterial stiffness induces progressive reduction of tensile strength, elongation and burst pressure with consequent drop of vessels breakpoint (10), that could be associated with vascular complications. Particularly, femoral artery stiffness could predispose to microlesions formation at TAVI device access, inducing vascular closure devices failure and vascular complications. Furthermore, vessel rigidity can be associated with a higher resistance during TAVI device delivery and increased probability of vessels injury (especially in presence of tortuosity and small artery diameters). Nowadays, there are no studies evaluating the relationship between arterial stiffness and TAVI vascular complications.

Aim The aim of this study is to evaluate the relationship between arterial stiffness and TAVI vascular complications, defining a new predictor of vascular complications in order to give more accurate information for procedures planning.

Endpoints The primary study endpoint is a composite of: any life-threatening, major or minor bleeding complication, or any major or minor vascular access complication according to VARC 3 criteria (6).

The secondary endpoints are: time to hemostasis, procedural length, in hospital/30 day any vascular complications, any bleedings, mortality, stroke/TIA, myocardial infarction and hospitalization, 1 year mortality, stroke/TIA, myocardial infarction, hospitalization and modified VCD failure, which was defined as failure of the VCD to achieve hemostasis within 5 min or requiring additional maneuvers (such as endovascular stenting, surgical techniques, balloon inflation or additional closure devices). 30-day PM implantation and FA insurgence/recurrence were also evaluated.

Methods

1) MEASUREMENTS OF ARTERIAL STIFFNESS Systemic and local arterial stiffness can be evaluated by different non-invasive methods. Pulse wave velocity (PWV) is the most widely used, non-invasive and accurate method for aortic stiffness evaluation. PWV is a strong predictor of cardiovascular worse outcome, now considered to be the gold standard arterial stiffness measurement (11,12). However, despite these advantages, PWV does not reflect the degree of arteriosclerosis in the local arterial wall, because it is an indirect measure of regional arterial stiffness and needs a special device scarcely available in hospital centers. To overcome PWV limitations, alternative methods have been proposed, in particular ultrasound methods are a useful tool for this purpose, allowing the direct visualization of the arterial wall, the measurement of blood flow using the Doppler technique and are available in vast majority of hospital centers (13,14).

1a. Echocardiographic Assessment of Aortic Pulse-Wave Velocity

Measurement of echocardiographic pulse wave velocity (PWV) needs the registration of doppler waveforms at two artery sites for the evaluation of transit time. The first acquisition should be in the distal aortic arch (T1:at level of left subclavian artery origin), the second one in the left distal external iliac artery (T2) and then the distance between artery sites should be calculated (D):

T1: time interval between the peak R wave on electrocardiography and the onset of PW Doppler signal of the descending thoracic aorta; T2: time interval between the peak R wave on electrocardiography and the onset of PW Doppler signal of the external iliac artery (EIA).

D: distance from the beginning site of the descending thoracic aorta (T1 evaluation point) to the EIA (T2 evaluation point) will be measured with Angio CT analysis.

Transit time (∆T): calculated as the difference between time from the QRS complex to the beginning of the EIA Doppler waveform (T2) and time from the QRS complex to the beginning of the distal aortic arch Doppler waveform (T1).

PWV: will be calculated as (T2-T1)/(D). Doppler sample volume will be set at 5.07 mm and the low-velocity filter will be reduced to get the beginning of the waveform adjacent to the baseline. 5 consecutive Doppler waveforms were recorded at a sweep speed of 100 mm/sec.

1b. Echocardiographic Assessment of Femoral stiffness

Femoral arterial stiffness indices were calculated according to the following formulas (13,15):

1. Arterial diameter change (mm)=SD-DD
2. Arterial strain=(SD-DD)/DD
3. Elastic modulus E(p)=(SBP-DBP)/strain
4. Arterial stiffness index ß=Ln (SBP/DBP)/strain (Ln: natural logarithm)
5. Arterial distensibility coefficient =(2×strain)/(SBP-DBP)

SD is systolic arterial diameter, DD is diastolic arterial diameter and SBP and DBP are brachial systolic and diastolic blood pressure, respectively. The use of brachial instead of local blood pressure (BP) may underestimate the predictive value of local stiffness due to BP amplification (i.e., the increase in BP along the arterial tree). The magnitude of amplification, however, tend to reduce with aging (14). Consequently, in elderly populations (13,16), local stiffness indices calculated with brachial or local PP may yield similar results. Stiffness index β, suggested by Hayashi et al. (17) provides a measurement of arterial stiffness independent of blood pressure at the time of measurement within the physiological blood pressure range (63-200 mmHg).

Measurement of femoral artery diameters will be acquired with linear probe only in patients with acceptable common femoral artery acoustic window and undergoing transfemoral-TAVI. M-Mode configuration with beam perpendicular to femoral artery (1 to 3 centimetres proximal from bifurcation) will be used for both SD and DD measurement.

2) PATIENTS ENROLLMENT

Consecutive patients will be enrolled before undergoing TAVI procedure:

Inclusion criteria

* Age ≥ 18 years
* Patients eligible for transfemoral TAVI. Exclusion criteria
* Conditions determining inadequate windows for evaluation of pulse wave doppler both at aortic arch and femoral artery level.
* CT scan not performed.
* Planned surgical access.

  3) DATA COLLECTION AND ANALYSIS Local database will be used for data collection and management. Ultrasound and CT scan acquisitions will be stored and evaluated offline using dedicated software (EchoPAC; GE Healthcare. Horos; Apple) by 2 expert investigators who will be blinded to clinical and laboratory data; in case of discordance, a consensus reading will be achieved with a third senior investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients eligible for transfemoral TAVI.

Exclusion Criteria:

* Conditions determining inadequate windows for evaluation of pulse wave doppler both at aortic arch and femoral artery level.
* CT scan not performed.
* Planned surgical access.

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: patients ≥ 75 years old with severe symptomatic aortic stenosis after Heart Team evaluation
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary study endpoint is a composite of: any life-threatening, major or minor bleeding complication, or any major or minor vascular access complication according to VARC 3 criteria (6). | 12 months
  The primary study endpoint is a composite of: any life-threatening, major or minor bleeding complication, or any major or minor vascular access complication according to VARC 3 criteria (6).

CONTACTS AND LOCATIONS:
Locations (1):
- A.O. Ordine Mauriziano, Torino, Italy

IPD SHARING:
Plan to Share IPD: Undecided